CLINICAL TRIAL: NCT05007067
Title: A Retrospective Study Evaluating Clinical and Radiographic Early Outcomes of Total Hip Arthroplasty With DELTA Multihole TT Acetabular Cup.
Brief Title: H-29 DELTA Multihole TT Study.
Status: Terminated | Type: Observational
Why Stopped: Lack of progress in fulfilling the Study activities, including the lack of enrollment of participants
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-29
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: DELTA Multihole TT — Advance articular destruction generated by primary degenerative or post-traumatic arthrosis or reumatoid arthritis; fracture or avascular necrosis; congenital or acquired deformity.

SUMMARY:
This study is aimed to provide a clinical and radiographic evaluation of 50 suitable subjects who underwent a complex primary or a revision Total Hip Arthroplasties with DELTA Multihole TT acetabular cup in 2019 onwards.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who underwent a Total Hip Arthroplasty with Delta Multihole TT acetabular cup, as per indications for use, in 2019 onwards
* Age ≥ 18 years old
* Subjects who have signed the written informed consent approved by the reference Ethics Committee (EC)
* Subjects able to comply with the protocol and to perform all scheduled follow-up visits

Exclusion Criteria:

* Male or female subjects who underwent a Total Hip Arthroplasty with Delta Multihole TT acetabular cup, but showed any of the contraindications reported in the Instruction for Use
* Age < 18 years old
* Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation including, but not limited to:

  1. significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery.
  2. neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device.
  3. known metabolic disorders leading to progressive bone deterioration.
* Hip replacement on the contralateral side performed within less than one year.
* Female subjects who are pregnant, nursing or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 50 consecutive subjects who underwent a THA with the DELTA Multihole TT acetabular cup. Patients are screened for enrolment into the study from a list of patients who had a surgery at the Samodzielny Publiczny Szpital Kliniczny im. Prof. Adama Grucy CMKP in 2019 onwards.
  Subjects who do not meet all the inclusion criteria or meet any exclusion criteria are excluded from study participation and should be considered as a Screening Failure.
  Subjects who meet all the inclusion criteria and none of the exclusion criteria and agree to participate in the study signing the Informed Consent Form are enrolled.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | Month 24
  The percentage of subjects showing a Harris Hip Score (HHS) equal or greater than "Good" (i.e. equal or greater than 80 points) at 2 years after the surgery.

SECONDARY OUTCOMES:
ROM measurement | Pre-operative - Month 24
  Functional changes in the ROM measurements from pre-operative (baseline) to 2 years after surgery.
VAS Pain | Pre-operative - Month 24
  Changes in the VAS Pain score from pre-operative (baseline) to 2 years after surgery.
Implant stability | Month 24
  Radiographic implant evaluation and stability assessment at 2 years after surgery.
Survival rate | Month 24
  Survival rate expressed with Kaplan-Meier estimator at 2 years after surgery
Safety assessment | Intra-operative, Week 2, Week 6, Month 6, Month 12, Month 24
  Incidence, type, and severity of all the Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Garlewicz, Principal Investigator — Samodzielny Publiczny Szpital Kliniczny im. Prof. Adama Grucy CMKP
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny im. Prof. Adama Grucy CMKP, Otwock, Poland

IPD SHARING:
Plan to Share IPD: No